CLINICAL TRIAL: NCT03232255
Title: Clinical Benefit of a Mouthrinse for the Treatment of Dentine Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100080
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Other: Mouthrinse (IQP-OLP-101)

INTERVENTIONS:
Other: Mouthrinse (IQP-OLP-101) — Rinse/gargle 10mL of Mouthrinse for 60 seconds after tooth brushing, twice a day.

SUMMARY:
This study is to evaluate the benefit and tolerability of a Mouthrinse (IQP-OLP-101) in the treatment of dentine hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. At least one hypersensitive tooth in everyday life after PAV 1 in-office visit
2. At least one hypersensitive tooth in everyday life with a regular pain perception of at least 2 times per week after PAV 1 visit
3. At least one tooth with dentine hypersensitivity to air stimulation → VAS ≥ 40mm at study entry
4. Any sensitive tooth showing exposure of cervical dentine (gum recession) and no acute signs of caries on the exposed root
5. For subjects entering the study at stage PAR-control: good healing of the periodontal surgery site, cause of pain must not be the result of the periodontal surgery
6. Age ≥ 18 years and ≤ 75 years
7. Willing and able to attend the on-study visits
8. Willing and able to understand and to follow the study procedures and instructions
9. Good oral hygiene throughout the study
10. Written informed consent before participation in the study
11. Subjects have undergone dental hygiene treatment immediately prior to study inclusion (except subjects entering the study at stage PAR-control)

Exclusion Criteria:

1. Hypersensitivity only due to sweets
2. Allergic reactions to any ingredients of InQpharm Mouthrinse e.g. chlorhexidine, zinc lactate
3. Professional desensitizing therapy during the previous 3 months; GLUMA (glutaraldehyde/hydroxyethyl methacrylate) desensitizer application within 6 months
4. Chronic systemic anti-inflammatory and analgesic medications
5. Systemic disorders causing or predisposing to dental (e.g. dry mouth, reflux, eating disorders, etc.)
6. Teeth or supporting structures with any other painful pathology or defect
7. Subject with poor health conditions
8. Concurrent participation in another clinical trial
9. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Change in dentine hypersensitivity | 28 days
  Assessed by subjects using VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Praxisklinik ORS, Fellbach, Germany

IPD SHARING:
Plan to Share IPD: No